CLINICAL TRIAL: NCT07197086
Title: Clinical and Treatment Determinant of Prognosis in Glioblastoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Afnan Mohamed Abd elaal, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: glioblastoma clinical &treat
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Adult patients (≥18 years) with histologically confirmed glioma (WHO grades 2-4)

SUMMARY:
Gliomas represent the most common primary malignant brain tumors in adults, with glioblastoma (WHO grade 4) being the most aggressive subtype. Despite advances in surgical techniques, radiotherapy, and chemotherapy, prognosis remains poor, particularly for high-grade gliomas. Maximal safe surgical resection is considered a cornerstone in the management of gliomas. Several studies suggest that a greater extent of resection (EOR) is associated with improved overall survival (OS) and progression-free survival (PFS), particularly in high-grade tumors. However, the benefit must be balanced against the risk of neurological deficits.

Postoperative chemoradiotherapy, particularly with temozolomide, has become the standard of care for high-grade gliomas. Despite this, the impact of EOR on outcomes in the context of adjuvant chemoradiotherapy remains a subject of ongoing investigation. This study aims to evaluate the prognostic significance of the extent of surgical resection in glioma patients who undergo postoperative chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with histologically confirmed glioma (WHO grades 2-4) Underwent neurosurgical resection (gross total, subtotal, or biopsy only) Received postoperative radiotherapy with or without concurrent and/or adjuvant temozolomide Available pre- and post-operative imaging for EOR assessment Complete medical records and follow-up data

Exclusion Criteria:

* Recurrent gliomas at presentation Incomplete treatment (e.g., abandonment, death before adjuvant therapy) Lack of imaging or follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with histologically confirmed glioma (WHO grades 2-4)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival (from surgery to death/last follow-up )which defined as the length of time from either the date of diagnosis or the start of treatment that patients diagnosed with the disease are still alive

IPD SHARING:
Plan to Share IPD: Yes